CLINICAL TRIAL: NCT06211413
Title: A Prospective Longitudinal Cohort Study of the Incidence of Hypertension and Arrhythmias in Patients Treated with Bruton's Tyrosine Kinase Inhibitors for Chronic Lymphocytic Leukemia Using Wearable Technology
Brief Title: Hypertension and Arrhythmias in CLL Patients Treated with BTK Inhibitors
Acronym: SENTINEL
Status: Enrolling by invitation | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 43421
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia; Atrial Fibrillation; Hypertension; Cardiotoxicity
Keywords: Acalabrutinib; Zanabrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Atrial Fibrillation; Hypertension; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Acalabrutinib and Zanabrutinib are highly effective drugs used to treat Chronic Lymphocytic Leukemia, but they are associated with high blood pressure and abnormal heart rhythms. SENTINEL is an observational study that will use wearable technology to monitor heart rhythm and blood pressures at home to better understand how frequently patients are experiencing high blood pressure and/or abnormal heart rhythms.

DETAILED DESCRIPTION:
Given the significant morbidity and mortality associated with hypertension and AF including stroke, systemic thromboembolism and heart failure, monitoring asymptomatic patients who are at high risk is an important area of investigation in the general population and is clearly an area of substantial need in the setting of BTK inhibitor use. Leveraging technology (including wearable and digital devices) to evaluate for the development of arrhythmias is an area of increasing focus in the field of cardiology and has led to various partnerships with technology companies including Apple, Google and Amazon. Several devices have shown promise in their ability to detect subclinical arrhythmias including patch and implantable recording devices, Smartwatches and digital sensors. Given the unmet need to better quantitate hypertension and arrhythmia burden in patients treated with BTK inhibitors, the investigators propose a study in which a SmartWatch, as well as at home blood pressure monitoring is used to monitor for the development of arrhythmias in either acalabrutinib- or zanubrutinib-treated CLL patients to better determine incidence and prevalence in a real world population. Based on these data, the investigators will be able to provide optimal treatment to patients while also ensuring accurate representation of hypertension and arrhythmia toxicity data which may translate into reductions in long term cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥22
* Initiation of BTK inhibitor (acalabrutinib or zanubrutinib) with or without other concurrent systemic therapy as front line or relapsed/refractory therapy for chronic lymphocytic leukemia, ordered by treating oncologist per standard of care
* Normal sinus rhythm at the time of consent
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Exclusion Criteria:

* Current use of a class IC or III antiarrhythmic medication
* AF or other arrhythmia at the time of consent
* Uncontrolled hypertension (≥140/90mmHg) at the time of consent
* Inability to provide informed consent
* Inability to wear a watch
* Arm circumference too small (< 9 in) or arm circumference too large (> 14.5in.) to use the QardioArm cuff
* Expected survival less than one year.
* Pregnancy at time of consent
* Lack of access to a personal Apple iPhone. If the patient does not have an Apple iPhone, but another member of the patient's household has an iPhone, the patient may still be enrolled as long as there is no other Apple Watch paired with the phone.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Lymphocytic Leukemia initiating therapy with acalabrutinib and/or zanabrutinib will be evaluated for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypertension | 6 months
  New onset or worsening hypertension recorded on home blood pressure monitoring

SECONDARY OUTCOMES:
Incidence of atrial or ventricular arrhythmias | 6 months
  Any episode of atrial or ventricular arrhythmias identified via wearable device monitoring
Incident episodes of major cardiovascular events | 6 months
  Incident episode of stroke/TIA, other thromboembolic events, heart failure, ischemic hear events
Bruton's Tyrosine Kinase inhibitor discontinuation | 6 months
  determination of the rate of Bruton's Tyrosine Kinase inhibitor discontinuation after development of arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fradley, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided